CLINICAL TRIAL: NCT02180984
Title: The Effects of Repetitive Transcranial Magnetic Stimulation in Obese Females With Binge Eating Disorder: a Protocol for a Double-blinded, Randomized, Sham-controlled Trial.
Brief Title: The Effects of Repetitive Transcranial Magnetic Stimulation in Obese People With BED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, ANGELICA CLAUDINO, Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 26164614.7.0000.5505; 26164614.7.0000.5505 (Other: CEP UNIFESP)
Record Dates: First submitted 2014-06-25; First posted 2014-07-03 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Binge Eating; Obesity
Keywords: Binge Eating; Obesity; TMS; Neuroimage; Neuromodulation; Biomarkers; Eating Disorders; Cognition; Endocrine; Hormones; BDNF; Inflammatory biomarkers
MeSH Terms: conditions — Bulimia; Obesity; Feeding and Eating Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Repetitive transcranial magnetic stimulation applied to people with binge eating disorder (real x sham stimulation) only (not for control groups without binge eating disorder)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only provider of the stimulation aware of allocation arm (real or sham)
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BED randomized to rTMS (Active Comparator): 30 obese individuals currently diagnosed with BED and meeting criteria for the study will be randomized to active rTMS treatment.
  Intervention: Neurosoft device targeting the left DLPFC (neuro-navigational method).
  Proposed schedule of treatment:
  20 sessions of neuronavigated rTMS, one session per day, 3 days/week over approximately 7 weeks. Focal rTMS will be performed using a Neurosoft device and a 'figure of eight' coil. Brainscience Neuronavigation will be used to guide the placement of the coil to the target PFC region using a template MRI for all participants. The coil will be placed at a 45° angle to the mid-sagittal line to induce a posterior to anterior current in the underlying neural tissue. For the real treatment condition, stimulation will target the left DLPFC at 110% of the resting motor threshold. Each session of 10 Hz stimulation will apply 1000 pulses to the left hemisphere, with a duty cycle of 5s on and 55s off, for a total stimulation time of 20 min.
  Interventions: Device: TMS
- Sham BED TMS (Sham Comparator): 30 obese individuals currently diagnosed with BED will be randomized to receive sham TMS treatment. Blinded to participants and study staff, except to the doctor applying the TMS treatment.
  Intervention: Neurosoft device targeting the left DLPFC (neuro-navigational method).
  Proposed schedule of treatment:
  20 sessions of neuronavigated rTMS, one session per day, 3 days/week over approximately 7 weeks. Focal rTMS will be performed using a Neurosoft device and a 'figure of eight' coil. Brainscience Neuronavigation will be used to guide the placement of the coil to the target PFC region using a template MRI for all participants. The coil will be placed at a 45° angle to the mid-sagittal line to induce a posterior to anterior current in the underlying neural tissue. Sham treatment condition, will follow the same protocol however no real TMS will be delivered.
  Interventions: Device: TMS
- Control (obese non BED) (No Intervention): 15 controls, obese but without a current or past diagnosis of BED will complete the baseline measurements only.
- Controls (normal weight) (No Intervention): 15 controls, normal weight and without a current or past diagnosis of BED will complete baseline measures only.

INTERVENTIONS:
Device: TMS — Transcranial Magnetic Stimulation has developed into a powerful tool that utilizes magnetic fluxes to non-invasively stimulate the human cortex. The technique involves placement of a small coil over the scalp; passing a rapidly alternating current through the coil wire, which produces a magnetic field that passes unimpeded through the scalp and bone, resulting in electrical stimulation of the cortex.
  Other Names: Repetitive Transcranial Magnetic Stimulation; Transcranial Magnetic Stimulation; rTMS
  Arms: BED randomized to rTMS; Sham BED TMS

SUMMARY:
The presence of binge eating (BE) is a core feature of bulimic syndromes. Binge eating disorder (BED) is a new category in DSM-5 highly associated with higher body mass index (BMI). The neural mechanisms that underlie BE are of great interest in order to improve treatment interventions. Brain mechanisms underlying drug and food craving are suggested to be similar. These mechanisms demonstrated hyperactivity in the orbitofrontal and anterior cingulate cortex and lack of regulatory influence from lateral prefrontal circuits. Several novel studies began to assess the potential benefits of brain stimulation in reducing craving and associated addictive behaviors with promising results. Previous findings testing a one-off session of repetitive transcranial magnetic stimulation (rTMS) in healthy women identified as strong cravers and individuals with bulimia nervosa or bulimic-type eating disorders reported reduction of food craving and BE, providing evidence to support a broader and deeper investigation of the benefits associated with rTMS. Importantly, the use of brain imaging studies contributes to the understanding of psychiatric disorders and underlying mechanisms being target by the rTMS intervention.

Objectives: The primary aim is to investigate the effects of rTMS over BE frequency. Secondary aims include the evaluation of the effects of rTMS on food craving, body weight, brain activity, cognition, general psychopathology, hormonal regulation and neurobiological markers. Methods: Sixty obese females with BED will be randomized to receive 20 sessions of rTMS (n=30) or placebo (n=30) scattered 3 days/week.

Expected Results: Primarily it is expected that rTMS intervention will decrease BE frequency. Consequently, body weight will be reduced. It is also expected that food craving be decreased, cognitive performance be enhanced, and neurobiological markers be improved.

DETAILED DESCRIPTION:
The primary aim is to investigate the effects of rTMS over BE frequency. Secondary aims include the evaluation of the effects of rTMS on food craving, body weight, brain activity, cognition, general psychopathology, hormonal regulation and neurobiological markers. Methods: Sixty obese females with BED will be randomized to receive 20 sessions of rTMS (n=30) or placebo (n=30) scattered 3 days/week.

Expected Results: Primarily it is expected that rTMS intervention will decrease BE frequency. Consequently, body weight will be reduced. It is also expected that food craving be decreased, cognitive performance be enhanced, and neurobiological markers be improved.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 55 years old
* Right handed
* Females
* BED diagnosis (EDE 16.0 - BED module) according to the DSM-5 criteria
* BMI ≥ 35kg/m2 and body weight ≤ 150kg
* Ability to write, read, and understand all elements of the study
* Safety laboratory blood work (fasting glucose, fasting glucose/insulin ratio, CBC, and TSH) within normal range
* Informed consent signed.

Exclusion Criteria:

* Past history of head or eye injury or epilepsy
* Body metallic implants, pacemaker, claustrophobia and any other contraindication to fMRI or rTMS;
* Current use of psychotropic drugs (except for antidepressants on a stable dose for at least one month)
* Current use of any anti-obesity drug (three months washout period for any other medication)
* Pregnancy or breastfeeding
* Diabetes Mellitus diagnosis
* Major psychiatric disorder requiring immediate treatment
* Substance dependence (SCID-I/P module for substance abuse and/or dependence applied for those who disclose substance use at checklist, following the DSM-5 criteria)
* Individuals currently receiving any psychological therapy for their eating disorder
* Cushing's and Turner's syndrome.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change in the number of binge eating episodes and craving. | Average of 2 months
  Weekly binge eating episodes frequency will be assessed by the medical doctor. The primary outcomes of this study are: (1) the change in the number of BE episodes before and after study treatment (number of BE episodes at baseline subtracted from the number of BE episodes at the end of treatment), as measured by participants recording of binge episodes in the food diary during the previous 15 days to the baseline visit (first rTMS session,T.3) to the end of treatment visit (T.23); (2) the change in "urge to eat" (craving) as measured in a 10 cm VAS (from T3 to T22).

SECONDARY OUTCOMES:
Change of food craving questionnaires (state and trait) scores | Average of 2 months (baseline and end of treatment)
  Food craving questionnaires scores will be analyzes at baseline and at the end of the treatment (approximately 2 months). Final scores for each of the participants will be subtracted from the baseline scores.
Change in Body Weight | Average of 2 months
  Reduction of baseline body weight (kg) at the end of the treatment (average of 2 months). The final weight will be subtracted from the baseline weight for each of the patients.
Binge eating episodes maintenance | 8 weeks follow up (after end of treatment)
  Weekly binge eating episodes frequency will be recorded by participants. Participants will asked to record date, time and description of binge eating episodes. The total number of episodes and frequency distribution for each of the groups will be analyzed.
Change of visual analogue scale scores | Average of 2 months (baseline and end of treatment)
  visual analogue scale scores will be analyzes at baseline and at the end of the treatment (approximately 2 months). Final scores for each of the participants will be subtracted from the baseline scores.

OTHER OUTCOMES:
Stroop test scores baseline difference. | Baseline
  Difference between groups of baseline Stroop test scores.
Assessment of adverse events and tolerability | Average of 2 months
  During the study participants will be asked if they are experiencing any of the expected adverse events or adverse events that are not expected. Number of expected and not expected adverse events will be recorded. Number of participants experiencing adverse events will be recorded. In addition participants will complete the tolerability scale at the end of each of TMS session and group mean score will be analyzed at the end of the treatment (average of 2 months).
Change in hormone levels | Average of 2 months
  Assessment of hormones (ghrelin (pg/mL), leptin (ng/mL), Peptide YY (pg/mL) and estrogen (pg/mL)), inflammatory biomarkers (PCR (mg/L), TNF-alpha(pg/mL), IL-6 (pg/mL), IL-10 (pg/mL)), anti-inflammatory biomarkers (adiponectin (µg/mL) and IL-2 (pg/mL)) and BDNF. Group mean baseline levels compared to group means at the end of treatment (average of 2 months).
Stroop test and fMRI | Baseline
  Stroop test performance during the fMRI will be analyzed between groups. Better inhibitory response and greater activation in response inhibition regions, such as DLPFC, will be analyzed to assess differences between groups (control and randomized).
Stroop test performance long term | Approximately 2 months
  Stroop test performance during the fMRI will be analyzed between groups. Better inhibitory response and greater activation in response inhibition regions, such as DLPFC, will be analyzed to assess differences between groups (placebo and sham).

CONTACTS AND LOCATIONS:
Overall Officials: Angélica M Claudino, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Universidade Federal de São Paulo (Federal University of Sao Paulo) (UNIFESP), São Paulo, Brazil

REFERENCES:
- [Background] Maranhao MF, Estella NM, Cury ME, Amigo VL, Picasso CM, Berberian A, Campbell I, Schmidt U, Claudino AM. The effects of repetitive transcranial magnetic stimulation in obese females with binge eating disorder: a protocol for a double-blinded, randomized, sham-controlled trial. BMC Psychiatry. 2015 Aug 12;15:194. doi: 10.1186/s12888-015-0569-8. PMID 26265452